CLINICAL TRIAL: NCT02764138
Title: Preventing Internalizing Psychopathology in Preadolescents Exposed to Chronic Stress
Brief Title: Preventing Internalizing in Preadolescents Exposed to Chronic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Martha E. Wadsworth, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R33MH107631 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-05-06 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Chronic Stress; Anxiety; Depression
Keywords: poverty; discrimination
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BaSICS Intervention (Experimental): Intervention = Building a String Identity and Coping Skills (BaSICS). Children randomized to participate in 16 twice weekly BaSICS intervention sessions. Children learn coping skills, identity development, and collective action as ways to buffer against chronic stress.
  These children also complete pre- and post-intervention assessments, as well as 3-month and 12-month follow-up assessments.
  Interventions: Behavioral: Building a Strong Identity and Coping Skills
- Comparison (No Intervention): These children complete assessments only--timed to coincide with the intervention groups' assessments: pre- and post-intervention assessments, as well as 3-month and 12-month follow-up assessments. No intervention.

INTERVENTIONS:
Behavioral: Building a Strong Identity and Coping Skills — Psychoeducational program to teach children coping skills, healthy identity development, and collective social action.
  Other Names: BaSICS
  Arms: BaSICS Intervention

SUMMARY:
Racial and socioeconomic disparities in physical and mental health problems are large, persistent, and severe; begin during childhood; and stem from in part damage to physiologic stress response systems caused by chronic stress. Discovery of ways to prevent and/or halt this progression of damage to a child's stress response system may offer new directions for combatting health disparities. This project will evaluate the efficacy of a new prevention program designed to teach preadolescent children effective ways for coping with chronic stress that will have direct effects on their physiologic stress response systems (hypothalamic-pituitary-adrenal axis) and ultimately prevent onset of anxiety, depression, and post-traumatic stress symptoms and disorders.

DETAILED DESCRIPTION:
Mental health problems disproportionately affect racial and ethnic minority populations, as well as populations that face chronic economic hardship. There is clear evidence that (1) the processes that lay the groundwork for mental health disparities is laid during childhood and (2) that damage to and dysregulation of the physiologic stress response is a powerful mechanism of the effects of chronic stress such as that associated with poverty on psychopathology. To contribute solutions to mental health disparities, interventions need to be capable of affecting the systems that confer the risk. Since the psychobiologic stress response system (e.g., hypothalamic-pituitary-adrenal axis; HPA) is a central mechanism linking health disparities to chronic stress, the stress response is a critical system to target. Improving children's ability to cope with stress and regulate their reactivity has the potential to break the cycle of damage, especially if the coping strategies and regulatory processes that we target have effects at the physiologic level. New evidence has emerged showing that different types of coping are evident at the level of the HPA-it is, therefore, time to evaluate whether a coping intervention designed for children facing chronic stress will both (a) improve children's ability to use primary and secondary control coping, and (b) have sustained effects at the physiologic level. The BaSICS intervention is designed to address core underlying mechanisms of risk and repair in the highly stressful context of poor, urban youths' lives.

Preadolescence is a crucial time during which children's ability to recognize stress and its causes matures, and repertoires for coping with stress grow in both size and complexity. In addition, preadolescence is a time of increased brain changes and growth in key self-regulatory organs and systems. Preadolescents are, therefore, at a ripe stage to benefit from coping-based prevention and the plasticity of this developmental period suggests that such changes have the potential to be long-lasting. BaSICS is designed to prevent the onset of anxiety, depression, and post-traumatic stress symptoms in preadolescent children facing chronic stress. Two mechanisms of action are targeted in this project. First, the project seeks to demonstrate that children facing chronic stress stemming from poverty, discrimination, and violence exposure can acquire and utilize new ways of coping that are adaptive in a wide variety of circumstances. Second, the project will examine the extent to which improved coping resulting from the intervention engages the physiologic intermediate mechanism of the HPA. Finally, the project aims to link changes in coping and the HPA to changes in internalizing symptoms that would signal prevention of the emergence of new or worsening of existing symptoms. Discovery of ways to prevent and/or halt this progression of damage to a child's stress response system that leads to psychopathology can offer new directions for combatting health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Child age 11 or 12 at intake
* Family income at or below 200% Federal Poverty Level
* Child speaks English
* Parent speaks English or Spanish

Exclusion Criteria:

* Intellectual disability
* Autism diagnosis
* Exceeds clinical cutoff for anxiety or depressive disorder

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2016-04; Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
HPA Reactivity Profile | Pre-post (3 months) and Pre-follow-up (6 and 12 months)
  Changes in levels of salivary cortisol across a 90 minute Trier Social Stress Test protocol

SECONDARY OUTCOMES:
Internalizing symptoms | Pre-follow-up (6 and 12 months)
  Reductions in total internalizing symptoms reported by parents on the CHild Behavior Checklist
Coping Skills Acquisition | pre-post (3 months) and Pre-follow-up (6 and 12 months)
  Changes in the number of coping skills that children can report during the Coping Skills interview protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Martha E Wadsworth, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Hamilton Health Center, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
National Data Archives